CLINICAL TRIAL: NCT05576792
Title: A 24-week, Open-label, Prospective, Single-arm Study Evaluating the Effectiveness and Safety of Lucentis® (Ranibizumab) 0.2mg in Retinopathy of Prematurity (ROP) Participants in China
Brief Title: A 24-week Study Evaluating the Effectiveness and Safety of Lucentis® 0.2mg in Retinopathy of Prematurity Participants in China
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRFB002H2403
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Retinopathy of Prematurity
Keywords: Retinopathy of Prematurity; ROP; NIS; China; ranibizumab
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- ranibizumab 0.2 mg: Intravitreal ranibizumab 0.2 mg for the treatment of ROP
  Interventions: Other: Ranibizumab

INTERVENTIONS:
Other: Ranibizumab — Prospective observational study. There is no treatment allocation. Patients prescribed with ranibizumab 0.2 mg in the commercial setting are eligible to enroll into this study.

SUMMARY:
This is a 24-week, multicenter, open-label, single-arm, observational, post approval commitment study, which is designed to collect effectiveness, safety and other clinical information of intravitreal ranibizumab 0.2 mg for the treatment of Retinopathy of Prematurity (ROP) participants in a real world clinical setting in mainland China.

DETAILED DESCRIPTION:
Eligible participants treated according to local routine clinical practice will be enrolled in the study upon signing an Informed Consent.

Participants will enter the study when they receive their first treatment and are followed up for 24 weeks. During the follow up period, participants could receive post-baseline treatment (i.e., ranibizumab or laser therapy) Patients will be treated according to the approved label and standard of care and as per Investigator judgement.

End of study will be defined as completion of the week 24 visit or premature withdrawal visit

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent from parent(s) or legal guardian(s), in compliance with local requirements
2. Male or female preterm infants with a birth weight of less than 1500 g
3. Bilateral ROP with 1 of the following retinal findings in each eye:

   * Zone I, stage 1+, 2+, 3 or 3+ disease, or
   * Zone II, stage 3+ disease, or
   * A-ROP

Exclusion Criteria:

1. Have a history of hypersensitivity (either the patient or the mother) to ranibizumab or any component of the ranibizumab formulation or to drugs of similar chemical classes
2. Have been previously exposed to any intravitreal or systemic anti-VEGF agent (either the patient or the mother during this child's pregnancy)
3. Have used (either the patient or the mother) other investigational drugs as part of another clinical study (other than vitamins and minerals) within 30 days or within 5 half-lives of the other investigational drug, whichever is longer
4. Have received any previous surgical or nonsurgical treatment for ROP (e.g., ablative laser therapy or cryotherapy, vitrectomy)
5. Participants who have contraindications according to locally approved ranibizumab label

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female preterm infants with confirmed diagnosis of bilateral ROP who require treatment in China
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with absence of active Retinopathy of Prematurity (ROP) and absence of unfavorable structural outcomes in both eyes during the observational period after starting study treatment. | Week 24
  To achieve this outcome, participants cannot fulfill any of the following criteria:
  * Require intervention for ROP in either eye at or before the 24week assessment visit with a treatment modality other than ranibizumab
  * Have active ROP in either eye at the 24week assessment visit
  * Have unfavorable structural outcomes in either eye at or before 24-week assessment visit

SECONDARY OUTCOMES:
Incidence of AEs | Up to 24 weeks
  Incidence of AEs will be collected
Assessment of length | Baseline, Week 12, and Week 24
  For the assessment of length the participant should be wearing minimal clothing (e.g., a clean diaper). Recumbent length in centimeters will be measured using an infantometer or according to local clinical practice.
Assessment of weight | Baseline, Week 12, and Week 24
  For the assessment of weight the participant should be wearing minimal clothing (e.g., a clean diaper). Body weight to the nearest gram will be measured using an electronic scale.
Assessment of head circumference | Baseline, Week 12, and Week 24
  For the assessment of head circumference the participant should be wearing minimal clothing (e.g., a clean diaper). The maximum occipitofrontal head circumference in centimeters will be measured using a tape measure.
Assessment of lower leg length | Baseline, Week 12, and Week 24
  For the assessment of lower leg length the participant should be wearing minimal clothing (e.g., a clean diaper).The lower leg length (knee-heel length) will be measured to the nearest 0.1 centimeter using a sliding caliper or according to local clinical practice. Measurements should always be done on the right side, unless a physical deformity affects the right side.
Time to intervention with a second modality for ROP or development of unfavorable structural outcome | Up to 24 weeks
  Time to intervention with a second modality for ROP or development of unfavorable structural outcome will be collected
Proportion of participants with re-treatment of ROP receiving any post-baseline intervention | 24 weeks
  Proportion of participants with re-treatment of ROP receiving any post-baseline intervention at or before 24 weeks
number of ranibizumab administrations needed in the treatment of participants with ROP | 24 weeks
  number of ranibizumab administrations needed in the treatment of participants with ROP will be collected
Full retinal vascularization in 12 clock hours | Week 24
  Full retinal vascularization in 12 clock hours at the 24-week assessment to evaluate fundus features of ranibizumab 0.2 mg in the treatment of ROP

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CRFB002H2403 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18264